CLINICAL TRIAL: NCT05266794
Title: A Novel Role of Alpha Lipoic Acid in Comparison With Selenium in Mitochondrial Resuscitation and miRNA-126 Expression in Hemodialysis Patients Randomized, Prospective, Controlled Study
Brief Title: A Novel Role of Alpha Lipoic Acid in Comparison With Selenium in Mitochondrial Resuscitation and miRNA-126 Expression in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MS 381/2018
Record Dates: First submitted 2022-02-18; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Antioxidative Stress; End Stage Renal Disease on Dialysis
Keywords: Oxidative stress; Antioxidants; mitochondrial function; CoQ10; miRNA-126; Hemodialysis
MeSH Terms: interventions — Thioctic Acid; Selenium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): 25 hemodialysis patients who received their routine therapy only.
- Selenium (Active Comparator): 23 hemodialysis patients who received Selenium 200µg once daily with their routine therapy just after the dialysis sessions for 3 months.
  Interventions: Drug: Selenium
- Alpha Lipoic acid (Active Comparator): 20 hemodialysispatients who received Alpha Lipoic acid (ALA) (Thiotex fort®) 600mg once daily with their routine therapy just after the dialysis sessions for 3 months.
  Interventions: Drug: Alpha lipoic acid

INTERVENTIONS:
Drug: Alpha lipoic acid — 20 patients who received Alpha Lipoic acid (ALA) (Thiotex fort®) 600mg once daily with their routine therapy just after the dialysis sessions for 3 months.
  Arms: Alpha Lipoic acid
Drug: Selenium — 23 patients who received Selenium 200µg once daily with their routine therapy just a
  Arms: Selenium

SUMMARY:
An Open labeled, Paralled, Randomized, Prospective, study was conducted on 60 patients who were randomized into 3 groups, 22, 20 and 18 patients in Control, Selenium and, Thiotacid groups respectively. Serum levels of ROS, CoQ10, and miRNA-126 were assessed at base line and after three months for all patients.

ELIGIBILITY:
Inclusion Criteria:

* prevalent hemodialysis patients

Exclusion Criteria:

* Patients with Inflammatory diseases, hepatic or respiratory diseases, smokers and alcoholics, were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change in miRNA-126 level | 3 months
  Fold expression
Change ROS level (ng/ml) | 3 months
  Using ELISA kit
Change in Co Q10 level (ng/ml) | 3 months
  Using ELISA kit

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided